CLINICAL TRIAL: NCT06911307
Title: Exploring the Effectiveness of Unpowered Negative Pressure Wound Therapy: a Randomized Controlled Trial
Brief Title: Exploring the Effectiveness of Unpowered Negative Pressure Wound Therapy
Acronym: NPWT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Collaborators: BenQ Materials Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID001; 000 (Other Grant/Funding Number: 000)
Record Dates: First submitted 2025-03-02; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-02

CONDITIONS: Chronic Wound; Acute Wound
Keywords: Negative Pressure Wound Therapy;; wound care; randomized controlled trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NPWT (Experimental): The NPWT group (experimental group) will include 80 participants. Wounds will be cleansed with sterile normal saline, followed by wound assessment and documentation. The Anscare SIMO Negative Pressure Wound Therapy (NPWT) System, a non-powered NPWT dressing, will then be applied.
  Interventions: Other: NPWT
- standard care group (Other): Thestandard care group will include 80 participants. Wounds will be cleansed with sterile normal saline and receive routine wound care, followed by wound assessment and documentation.
  Interventions: Other: standard care group

INTERVENTIONS:
Other: standard care group — The standard care (SC) group will also include 80 participants. Wounds will be cleansed with sterile normal saline and managed using conventional wound care techniques. Participants will undergo regular postoperative follow-ups to assess wound healing progression and secondary outcome measures.
  Arms: standard care group
Other: NPWT — The NPWT group will also include 80 participants. Wounds will be cleansed with sterile normal saline and coverd the SIMO NPWT dressing. Participants will undergo regular postoperative follow-ups to assess wound healing progression and secondary outcome measures.
  Arms: NPWT

SUMMARY:
The aim of this study is to investigate the effectiveness of Non-powered Negative Pressure Wound Therapy (NPWT) on the healing of abdominal surgical wounds. It is designed as a randomized controlled trial with an experimental group (using NPWT) and a control group (conventional wound care). The study aims to recruit 160 participants: 80 with acute wounds and 80 with chronic wounds. Participants will be randomly assigned to either the experimental group (40 acute wounds, 40 chronic wounds) or the control group (40 acute wounds, 40 chronic wounds). The study will assess wound healing rates and speed, quality of life, self-perceived health status, pain levels, complications, and wound care costs using indicators. Effectiveness will be analyzed using Generalized Estimating Equations (GEE). The study anticipates that results will contribute to evaluating the effects of Non-powered NPWT on wound healing, quality of life, pain, and cost-effectiveness in patients with acute and chronic wounds.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with acute wounds (wound duration <4 weeks) or chronic wounds (wound duration ≥4 weeks).
2. Wound depth <2 cm.
3. Age ≥18 years.
4. Patients who have been evaluated and approved for participation by their attending physician.

Exclusion Criteria:

1. Patients with unstable vital signs.
2. Presence of ischemia in the wound or surrounding tissues.
3. Fragile skin around the wound.
4. Severe wound infection or necrotic tissue.
5. Wound size >10 × 20 cm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
wound healing | 90days
  1. Wound size will be measured before and after the intervention, using a ruler and photographic records.
  2. The occurrence and time of healing events will be documented. The modified TIME-H score will be used as the evaluation tool. This scoring system includes four main indicators: T (Tissue)、I (Infection)、M (Moisture)、E (Edge)、H (Healing).

SECONDARY OUTCOMES:
Pain Assessment | 90days
  Pain quality will be evaluated before and after the intervention using the Numeric Rating Scale (NRS), where 0 represents no pain and 10 represents the worst possible pain. The pain index will be recorded, and the type, frequency, and dosage of pain medication used during the enrollment process will be documented.
Wound-related Quality of Life | 90days
  The Wound-QoL-17 questionnaire will be used before and after the intervention to assess the quality of life related to the wound. The Wound-QoL-17 consists of 17 items across three domains: Physical, Psychological, and Daily Life. The responses are based on a 5-point Likert scale, where a higher score indicates poorer quality of life. The Cronbach's α for the original Wound-QoL-17 ranges from 0.71 to 0.916, while for the Chinese version, it ranges from 0.71 to 0.93, indicating good internal consistency (Cronbach's alpha).
Self-reported Health Status | 90days
  The PHQ-9 (Patient Health Questionnaire-9) will be used before and after the intervention to screen for and track symptoms of depression. The PHQ-9 consists of 9 questions, each evaluating depressive symptoms over the past two weeks. Responses are rated from "not at all" to "nearly every day", with the frequency of responses used to assess the severity of depression.
Length of Hospital Stay for wound treatment | 90days
  The number of days participants are hospitalized during the enrollment and follow-up periods due to their wound will be recorded.
Cost Analysis | 90days
  The cost of wound treatment during the enrollment and follow-up periods will be assessed, including: Direct wound dressing costs、Wound care technique fees、Wound-related surgery costs、Wound-related medication usage、Outpatient follow-up or dressing change costs.
Complications and Adverse Events | 90days
  The following will be monitored: Surgical Site Infection (SSI)、Wound dehiscence、Allergic reactions、Wound infection、Hematoma、Inflammation、Bleeding.
Adhesion Issues for Dressing | 90days
  This will include incidents of unintended dressing detachment, skin tear during dressing removal, and the methods of enhanced dressing fixation during treatment.
Mortality Events | 90days
  The cause and time of death for participants during the enrollment and follow-up periods will be recorded.

IPD SHARING:
Plan to Share IPD: No
The plan is not public yet.